CLINICAL TRIAL: NCT04023331
Title: 67Cu-SARTATE™ Peptide Receptor Radionuclide Therapy Administered to Pediatric Patients With High-Risk Neuroblastoma: A Multi-center, Dose-escalation, Open-label, Non-randomized, Phase 1-2a Theranostic Clinical Trial
Brief Title: 67Cu-SARTATE™ Peptide Receptor Radionuclide Therapy Administered to Pediatric Patients With High-Risk, Relapsed, Refractory Neuroblastoma
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: Clarity Pharmaceuticals Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CL04
Record Dates: First submitted 2019-07-14; First posted 2019-07-17 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Neuroblastoma; Relapsed Neuroblastoma; Refractory Neuroblastoma
MeSH Terms: conditions — Neuroblastoma | interventions — 64Cu-SARTATE

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- 67Cu-SARTATE (Experimental): 64Cu-SARTATE - patients will receive a bolus injection of 64Cu-SARTATE during screening, and following each 67Cu-SARTATE Therapy Cycle, at a rate of 2.0 MBq/kg.
  67Cu-SARTATE - In the dose escalation phase, patients will receive a single administration of 67Cu-SARTATE as an IV infusion (dose will be determined based on cohort allocation). In the expansion phase, patients will receive at least 2 administrations of 67Cu-SARTATE at the MTD/MFD level as a slow IV infusion.
  Participants in either phase of the study that demonstrate therapeutic benefit following treatment with 67Cu-SARTATE at any dose may be offered additional Therapy Cycles (each participant may receive a maximum of 4 Therapy Cycles in total).
  Interventions: Drug: 67Cu-SARTATE; Drug: 64Cu-SARTATE

INTERVENTIONS:
Drug: 67Cu-SARTATE — 67Cu-labelled MeCOSar-Tyr3-octreotate
  Other Names: Cu-67 SARTATE, copper 67 SARTATE
Drug: 64Cu-SARTATE — 64Cu-labelled MeCOSar-Tyr3-octreotate
  Other Names: Cu-64 SARTATE, copper 64 SARTATE

SUMMARY:
The aim of this study is to evaluate the safety and efficacy of 67Cu-SARTATE in pediatric patients with high-risk neuroblastoma.

DETAILED DESCRIPTION:
This is an 'adaptive trial'. The trial design uses the accumulating data from the ongoing trial to modify aspects of the trial (e.g. dose, number of treatments). The trial is also a 'personalised trial' as the interval between treatments and number of treatments is determined for each patient individually.

This study is to be conducted in 2 phases, a dose escalation phase and a cohort expansion phase.

Dose escalation will be completed using a modified 3+3 study design with up to 7 Cohorts of increasing doses in MBq/kg. Pre-defined Dose Limiting Toxicities will be monitored for 6 weeks post administration of 1 therapy cycle of 67Cu-SARTATE.

Participants who demonstrate therapeutic benefit (defined as non progression as assessed by the Investigator using the International Neuroblastoma Response Criteria (INRC) guidelines) may be offered additional Therapy Cycles (each participant may receive a maximum of 4 Therapy Cycles in total).

Cohort expansion will commence once either the Maximum Tolerated Dose (MTD) or the Maximum Feasible Dose (MFD) for a single administration of 67Cu-SARTATE is established, or Cohort 7 has been completed. The study will be expanded to enroll an additional 10 subjects who will receive at least 2 therapy cycles of 67Cu-SARTATE at the MTD/MFD dose level. Participants who demonstrate therapeutic benefit (defined as non progression as assessed by the Investigator using the INRC guidelines) may be offered additional Therapy Cycles (each participant may receive a maximum of 4 Therapy Cycles in total).

The study also includes a long-term follow-up period to 36 months following the first dose of 67Cu-SARTATE, although in person study visits are not required.

ELIGIBILITY:
Inclusion Criteria:

1. Participant is able and willing to provide informed consent (≥18 years), or informed consent is obtained by the parent or legal guardian for minor participants, with the minor providing age appropriate assent, according to local law and regulations;
2. Life expectancy ≥ 12 weeks for patients in the Dose Escalation Phase or ≥ 4 months for patients in the Cohort Expansion Phase;
3. Known high-risk neuroblastoma OR previously intermediate-risk neuroblastoma that has relapsed or progressed to high-risk, with failure to achieve complete response with standard therapy (defined as at least 4 cycles of aggressive multi-drug induction chemotherapy with or without radiation and surgery, or according to a standard high-risk treatment/neuroblastoma protocol), OR who are medically ineligible to receive standard treatment OR who are intolerant to standard treatment;
4. Adequate recovery from acute toxic effects of any prior therapy, as deemed by the Investigator or treating Sub-Investigator;
5. Adequate liver function as defined by the following laboratory values obtained within 28 days prior to administration of 64Cu-SARTATE: Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) < 3.0 x upper limit of normal (ULN);
6. Adequate renal function;
7. Adequate laboratory parameters: Absolute neutrophil count > 1.0 x 10 9/L; Platelet count > 50 x 10 9/L; Total bilirubin <1.5 x ULN;
8. Karnofsky or Lansky performance status ≥50;
9. All participants must have a hematopoietic stem cell product available (minimum CD34+ cell dose is ≥2 x 10 6 cells/kg);
10. Sexually active participants of reproductive potential must practice an effective method of birth control while participating on this study, to avoid possible damage to the fetus. Abstinence is considered acceptable;
11. 64Cu-SARTATE uptake on the 4 hour scan (SUVmax) of any lesion equal to or higher than that of the liver in order to move on to the therapy phase of the study.

Exclusion Criteria:

1. Participants with disease of any major organ system that would compromise their ability to tolerate therapy, as deemed by the Investigator or treating Sub-Investigator;
2. Participants with intracranial tumor affecting the brain parenchyma that has not been previously treated at the time of study enrolment;
3. Any other active malignancy, or a history of prior malignancy within the past 3 years;
4. History of cardiac failure as evidenced by: dyspnea at rest, exercise intolerance, oxygen requirement, clinically significant cardiac dysfunction;
5. Planned administration of chemotherapy, anti-cancer cytokine therapy, immunotherapy or radiotherapy within 2 weeks prior to the administration of 64Cu-SARTATE;
6. Administration of therapeutic dose of 131I-MIBG within 8 weeks prior to the administration of 64Cu-SARTATE;
7. External beam radiation therapy (EBRT) to both kidneys or a single functioning kidney within 12 months prior to the administration of 64Cu-SARTATE;
8. Administration of any investigational agents within 21 days prior to administration of 64Cu-SARTATE;
9. Treatment with long acting somatostatin analogues (administered within 28 days prior to the administration of 64Cu-SARTATE), or short acting somatostatin analogues (administered within 24 hours prior to the administration of 64Cu-SARTATE);
10. Known sensitivity or allergy to somatostatin analogues;
11. Previous peptide receptor radionuclide therapy (PRRT);
12. Female participants who are pregnant or lactating;
13. Participants who are on hemodialysis;
14. QTcF interval ≥ 0.45 seconds as measured by Screening ECG;
15. Participants with uncontrolled infection(s);
16. Any medical condition which the Investigator feels may interfere with the procedures or evaluations of the study;
17. Participants 12 months and younger will be excluded from cohorts where the planned single or cumulative administered activity is modelled to deliver a radiation dose to the marrow that exceeds 2 Gy.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2020-08-18 (Actual); Primary Completion 2025-01-24 (Actual); Study Completion 2025-03-25 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD)/Maximum Feasible Dose (MFD) of 67Cu-SARTATE | 6 weeks
  MDT/MFD as determined by cohort observations of Dose Limiting Toxicities
Safety and tolerability of 67Cu-SARTATE using Common Terminology Criteria for Adverse Events (CTCAE) | Up to 36 months
  Safety will be assessed via vital signs, pathology tests (hematology, biochemistry, urinalysis, coagulation), physical examinations, electrocardiograms (ECGs) and spontaneous adverse event (AE) reporting.
Safety and tolerability of 64Cu-SARTATE using CTCAE | Up to 36 months
  Safety will be assessed via vital signs, pathology tests (hematology, biochemistry, urinalysis, coagulation), physical examinations, ECGs and spontaneous AE reporting.
Overall response rate | Up to 12 months
  As assessed by international neuroblastoma response criteria (INRC).
Best response | 6 to 8 weeks post final therapy
  As assessed by international neuroblastoma response criteria (INRC).

CONTACTS AND LOCATIONS:
Locations (8):
- United States (8):
  - Phoenix Children's Hospital, Phoenix, Arizona
  - Washington University School of Medicine, St Louis, Missouri
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Cincinnati Children's Hospital Medical Centre, Cincinnati, Ohio
  - Medical University of South Carolina, Charleston, South Carolina
  - University of Texas Southwestern Medical Centre, Dallas, Texas
  - MD Anderson Cancer Center, Houston, Texas
  - University of Wisconsin, Madison, Wisconsin